CLINICAL TRIAL: NCT01002755
Title: Combination of Lenalidomide and Ofatumumab in Patients With Previously Treated Chronic Lymphocytic Leukemia and Small Lymphocytic Lymphoma (CLL/SLL)
Brief Title: Lenalidomide and Ofatumumab in Treating Participants With Previously Treated Chronic Lymphocytic Leukemia or Small Lymphocytic Lymphoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2009-0283; NCI-2018-01829 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 2009-0283 (Other: M D Anderson Cancer Center); P30CA016672 (NIH)
Record Dates: First submitted 2009-10-26; First posted 2009-10-27 (Estimated); Results first posted 2019-05-07 (Actual); Last update posted 2019-05-07 (Actual); Status verified 2019-04

CONDITIONS: Chronic Lymphocytic Leukemia; Fatigue; Fever; Hypogammaglobulinemia; Lymphadenopathy; Lymphocytosis; Night Sweats; Paraproteinemia; Small Lymphocytic Lymphoma; Thrombocytopenia
MeSH Terms: conditions — Leukemia, Lymphocytic, Chronic, B-Cell; Fatigue; Fever; Agammaglobulinemia; Lymphadenopathy; Lymphocytosis; Paraproteinemias; Thrombocytopenia | interventions — Lenalidomide; ofatumumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment (lenalidomide, ofatumumab) (Experimental): Participants receive ofatumumab IV over 4 hours on days 1, 8, 15, and 22 of course 1, day 1 of courses 2-6, and day 1 of every even course beginning course 8. Beginning day 9 of course 1, participants also receive lenalidomide PO daily. Courses repeat every 28 days for up to 2 years in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Lenalidomide; Biological: Ofatumumab

INTERVENTIONS:
Drug: Lenalidomide — Given PO
  Other Names: CC-5013; CC5013; CDC 501; Revlimid
Biological: Ofatumumab — Given IV
  Other Names: Arzerra; GSK1841157; HuMax-CD20; HuMax-CD20, 2F2

SUMMARY:
This phase II trial studies how well lenalidomide and ofatumumab work in treating participants with previously treated chronic lymphocytic leukemia or small lymphocytic lymphoma. Drugs used in chemotherapy, such as lenalidomide, work in different ways to stop the growth of tumor cells, either by killing the cells, by stopping them from dividing, or by stopping them from spreading. Monoclonal antibodies, such as ofatumumab, may interfere with the ability of tumor cells to grow and spread. Giving lenalidomide and ofatumumab may work better in treating participants with chronic lymphocytic leukemia or small lymphocytic lymphoma

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To evaluate efficacy and tolerability of the combination of ofatumumab and lenalidomide in patients with recurrent chronic lymphocytic leukemia (CLL).

OUTLINE:

Participants receive ofatumumab intravenously (IV) over 4 hours on days 1, 8, 15, and 22 of course 1, day 1 of courses 2-6, and day 1 of every even course beginning course 8. Beginning day 9 of course 1, participants also receive lenalidomide orally (PO) daily. Courses repeat every 28 days for up to 2 years in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, participants are followed up at 6 months, then every 3 months thereafter.

ELIGIBILITY:
Inclusion Criteria:

* Understand and voluntarily sign an informed consent
* Patients with CLL or small lymphocytic lymphoma (SLL) with active disease: B-CLL Rai III-IV or earlier stage disease with evidence of "active disease" as defined by the National Cancer Institute (NCI)-sponsored working group 1) weight loss of > 10% in prior 6 months, 2) extreme fatigue, 3) fever or night sweats without evidence of infection, 4) worsening anemia or thrombocytopenia, 5) progressive lymphocytosis with a rapid lymphocyte doubling time, 6) marked hypogammaglobulinemia or paraproteinemia, 7) lymphadenopathy > 5 cm in diameter
* Prior treatment with purine analog based chemotherapy or chemoimmunotherapy
* Platelet count > or = to 30,000 mm^3
* Eastern Cooperative Oncology Group (ECOG)/World Health Organization (WHO) performance status of 0-2
* Creatinine clearance > 30 ml/min (calculated by 24 hours urine collection) or a glomerular filtration rate (GFR) > 30 ml/min estimated using the Cockcroft-Gault equation
* Total bilirubin less or equal to 2 mg/dl
* Alanine aminotransferase (ALT) less or equal to two times the upper limit of normal
* Disease free of prior malignancies for 3 years with exception of currently treated basal cell, squamous cell carcinoma of the skin, or carcinoma "in situ" of the cervix or breast. Patients with malignancies with indolent behavior such as prostate cancer treated with radiation or surgery can be enrolled in the study as long as they have a reasonable expectation to have been cured with the treatment modality received
* Females of childbearing potential (FCBP) must have a negative serum or urine pregnancy test with a sensitivity of at least 50 mIU/mL within 10-14 days prior to starting lenalidomide and again within 24 hours prior to prescribing lenalidomide (prescriptions must be filled within 7 days) and prior to first ofatumumab administration and must either commit to continued abstinence from heterosexual intercourse or begin two acceptable methods of birth control, one highly effective method and one additional effective method at the same time, at least 28 days before she starts taking lenalidomide and continue it for 6 months after therapy has been completed. FCBP must also agree to ongoing pregnancy testing. Men must agree to use a latex condom during sexual contact with a FCBP even if they have had a successful vasectomy. All study participants must be registered into the mandatory RevAssist program, and be willing and able to comply with the requirements of RevAssist

Exclusion Criteria:

* Known sensitivity to lenalidomide, other thalidomide derivatives or ofatumumab
* Documented prolymphocytic leukemia (prolymphocytes more than 55% in the blood)
* Known positivity for human immunodeficiency virus (HIV) or active hepatitis B or C. Positive serology for hepatitis B (HB) defined as a positive test for hepatitis B surface antigen (HBsAg). In addition, if negative for HBsAg positive but HBcAb positive regardless of HBsAg status, a HB deoxyribonucleic acid (DNA) test will be performed and if positive the subject will be excluded
* Pregnant or breast feeding females. Women of childbearing potential must have a negative pregnancy test at screening. Male subjects unable or unwilling to use adequate contraception methods from study start to one year after the last dose of protocol therapy
* Chronic or current infectious disease requiring systemic antibiotics, antifungal, or antiviral treatment such as, but not limited to, chronic renal infection, chronic chest infection with bronchiectasis and tuberculosis. History of tuberculosis treated within the last five years or recent exposure to tuberculosis
* Any serious medical condition, laboratory abnormality, or psychiatric illness that places the subject at unacceptable risk if he/she were to participate in the study
* Patients with a recent history of deep vein thrombosis (DVT) or pulmonary embolus (PE), in the six months prior to enrollment are not eligible for this study
* Treatment with any known non-marketed drug substance or experimental therapy within 5 terminal half lives or 4 weeks prior to enrollment, whichever is longer, or currently participating in any other interventional clinical study
* Prior treatment with other monoclonal antibodies within 4 weeks prior to enrollment

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2010-01-19 (Actual); Primary Completion 2018-01-31 (Actual); Study Completion 2018-01-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Alessandra Ferrajoli, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- M D Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- [Derived] Takahashi K, Hu B, Wang F, Yan Y, Kim E, Vitale C, Patel KP, Strati P, Gumbs C, Little L, Tippen S, Song X, Zhang J, Jain N, Thompson P, Garcia-Manero G, Kantarjian H, Estrov Z, Do KA, Keating M, Burger JA, Wierda WG, Futreal PA, Ferrajoli A. Clinical implications of cancer gene mutations in patients with chronic lymphocytic leukemia treated with lenalidomide. Blood. 2018 Apr 19;131(16):1820-1832. doi: 10.1182/blood-2017-11-817296. Epub 2018 Jan 22. PMID 29358183
- See also: MD Anderson Cancer Center Website — http://www.mdanderson.org

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Treatment (Lenalidomide, Ofatumumab)
Started | 36
Completed | 36
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Treatment (Lenalidomide, Ofatumumab)
Number analyzed (Participants) | 36
Age, Continuous [Median (Full Range); unit: years] | 64 [34 to 82]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9
  Male | 27
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 3
  White | 32
  More than one race | 0
  Unknown or Not Reported | 1
Region of Enrollment [Number; unit: participants]
  United States | 36

OUTCOME MEASURES:

1. Primary Outcome: Overall Response Rate
Description: A Simon's two-stage minmax design will be used. Includes complete remission (CR) and partial remission (PR). Complete Response Requires the absence of disease signs and symptoms, and normalization of Peripheral blood and bone marrow. Partial Response it at lease a 50% reduction in disease signs and symptoms and normalization of peripheral blood.
Time Frame: Up to 8 years
Population: Two participants were not evaluable for response.
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment (Lenalidomide, Ofatumumab)
Number analyzed (Participants) | 34
Participants | 24

2. Secondary Outcome: Number of Participants With Tolerance of the Medication Combination
Description: Incidence of grade 3 and 4 non-hematological toxicity in more than 50 percent of the participants. Will be monitored based on the Bayesian model (beta-binomial).
Time Frame: Up to 8 years
Measure: Number; unit: participants
Arm/Group | Treatment (Lenalidomide, Ofatumumab)
Number analyzed (Participants) | 36
participants | 0

3. Secondary Outcome: Progression Free Survival
Description: The time from the start of therapy to death, disease progression, or the initiation of the next therapy. Disease progression is the loss of response or transformation to a more aggressive histology.
Time Frame: Up to 8 years
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Treatment (Lenalidomide, Ofatumumab)
Number analyzed (Participants) | 34
months | 16 [2 to 26]

ADVERSE EVENTS:
Time Frame: 1 year
Arm/Group | Treatment (Lenalidomide, Ofatumumab)
All-Cause Mortality (participants affected / at risk) | 0/36
Serious Adverse Events (participants affected / at risk) | 13/36
Other Adverse Events (participants affected / at risk) | 33/36
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (Lenalidomide, Ofatumumab) (N=36)
Adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Appendectomy (Surgical and medical procedures) | 1 (1)
Atrial Fibrillation (Cardiac disorders) | 1 (2)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 2 (4)
Fatigue (General disorders) | 1 (1)
Fever (General disorders) | 3 (4)
Hernia repair (Surgical and medical procedures) | 1 (1)
Infection (Infections and infestations) | 3 (3)
Meninogencephalitis (Infections and infestations) | 1 (1)
Neutropenic Fever (Infections and infestations) | 1 (2)
Pulmonary Embolism (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Thrombosis (Blood and lymphatic system disorders) | 2 (2)
Weakness (General disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (Lenalidomide, Ofatumumab) (N=36)
Acne (Skin and subcutaneous tissue disorders) | 3 (3)
Allergic Drug Reaction (Investigations) | 8 (11)
Anemia (Blood and lymphatic system disorders) | 10 (10)
Constipation (Gastrointestinal disorders) | 12 (12)
Cough (General disorders) | 8 (8)
Dermatology/Skin (Skin and subcutaneous tissue disorders) | 2 (2)
Diarrhea (Gastrointestinal disorders) | 15 (15)
Distention/Bloating (Gastrointestinal disorders) | 2 (2)
Dry eye (Eye disorders) | 2 (2)
Dry Skin (Skin and subcutaneous tissue disorders) | 2 (2)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 5 (5)
Edema Limb (Blood and lymphatic system disorders) | 2 (2)
Fatigue (General disorders) | 16 (16)
Fever (General disorders) | 14 (14)
Hyperglycemia (Metabolism and nutrition disorders) | 2 (2)
Hypomagnesemia (Metabolism and nutrition disorders) | 2 (2)
Infection (Infections and infestations) | 20 (20)
Insomnia (Nervous system disorders) | 2 (2)
Muscle Weakness (Musculoskeletal and connective tissue disorders) | 2 (2)
Nausea (Gastrointestinal disorders) | 9 (9)
Neurology other (Nervous system disorders) | 5 (5)
Neutropenia (Blood and lymphatic system disorders) | 23 (23)
Pain (General disorders) | 16 (16)
Pleural Effusion (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Pruritis (Skin and subcutaneous tissue disorders) | 6 (6)
Pulmonary Other (Respiratory, thoracic and mediastinal disorders) | 3 (3)
Rash/desquamation (Skin and subcutaneous tissue disorders) | 2 (2)
Sweating (General disorders) | 2 (2)
Thrombocytopenia (Blood and lymphatic system disorders) | 12 (12)
Tumor Flare (Immune system disorders) | 7 (7)
Vomiting (Gastrointestinal disorders) | 3 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2010-08-17): https://cdn.clinicaltrials.gov/large-docs/55/NCT01002755/Prot_SAP_000.pdf